CLINICAL TRIAL: NCT03733587
Title: A Phase 1b Study of GX-I7 in Combination With Cyclophosphamide in Patients With Metastatic or Recurrent Solid Tumors
Brief Title: GX-I7 With Cyclophosphamide in Patients With Metastatic or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GX-I7-CA-005
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — efineptakin alfa; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide and GX-I7 (Experimental): Cyclophosphamide and determined dose of GX-I7 of each cycle
  Interventions: Drug: GX-I7; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: GX-I7 — GX-I7 25mg/ml/vial
Drug: Cyclophosphamide — Cyclophosphamide 500mg/vial
  Other Names: Endoxan

SUMMARY:
This is a Phase 1b study to explore the safety and efficacy of GX-I7 in combination with CPA in patients with metastatic or recurrent solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1b study to explore the safety and efficacy of GX-I7 in combination with CPA in patients with metastatic or recurrent solid tumors.

This is 4 dose levels and increase dose level after confirm DLT of the previous dose.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of solid tumor, for which no standard therapy exists or is available any longer.
* Aged ≥19 years(Korean age).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy ≥12 weeks.
* Adequate hematological and end organ function defined by the following
* laboratory results obtained within 14 days prior to Cycle 1 Day 1 (C1D1)
* Female subjects of childbearing potential (including a female who has undergone tubal ligation) requires a negative serum pregnancy test performed within 14 days prior to C1D1.
* Have an evaluable lesion(s) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Subjects to be enrolled in the Phase 2a stage must be able to provide pre-treatment tissue biopsy or archival tissue and must have a tumor lesion.
* Providing the signed informed consent form (ICF).

Exclusion Criteria:

* Unable to adhere to the study procedures and follow-up procedures.
* Pregnant or lactating subjects.
* Have alcoholic or other hepatitis, liver cirrhosis, or genetic liver disease.
* Have uncontrolled type 2 diabetes mellitus.
* Have history of a major surgery within 28 days prior to C1D1 or are anticipated to require a major surgery during the study.
* Have an evidence of severe or uncontrolled systemic disease, uncontrolled hypertension.
* Have received any other investigational or approved anticancer therapy within 3 weeks prior to C1D1.
* With a positive result of human immunodeficiency virus (HIV) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Incidence of DLT | within cycle 1(28days)
  Incidence of nature of DLTs
Incidence and characteristics of AE | up to 24 months
  Incidence, nature and severity of adverse events graded according to NCI CTCAEv4.03
ORR | up to 6 months
  ORR defined as complete response (CR) or partial response (PR) per RECIST v1.1

SECONDARY OUTCOMES:
Incidence of ADAs | up to 24 months
  Incidence of anti-drug antibodies (ADAs) during the study
concentration of GX-I7 | up to cycle 3 day 1(approximately 8 weeks)
  Serum concentration of GX-I7 at specified timepoints for the Area under the concentration time-curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Minkyu Heo, Study Director — Genexine_clinical team
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No